CLINICAL TRIAL: NCT03454087
Title: Study of Early Enteral Dextrose in Sepsis
Acronym: SEEDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Faraaz Shah, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO17010532; 5K23GM122069 (NIH)
Record Dates: First submitted 2018-02-19; First posted 2018-03-05 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Sepsis
Keywords: enteral nutrition; inflammation; incretin hormones; microbiome
MeSH Terms: conditions — Sepsis; Inflammation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a blinded 1:1 fashion to receive either a low level enteral infusion of dextrose solution (intervention group) or an enteral infusion of free water (placebo group)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Infusion solutions will be prepared by pharmacy services at the local institution but participants, investigators, care providers, and outcomes assessors will be blinded to group allocation until the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enteral Dextrose Infusion (Experimental): Critically-ill participants with sepsis enrolled in the interventional arm will receive a 24-hour infusion of dextrose solution by the enteral route to be initiated via an existing nasogastric or orogastric tube within the first 48 hours of meeting sepsis criteria.
  Interventions: Other: Enteral Dextrose Infusion
- Placebo (Placebo Comparator): Critically-ill participants with sepsis in the placebo arm will receive a 24-hour enteral free water infusion via an existing orogastric or nasogastric tube within 48 hours of meeting sepsis criteria.
  Interventions: Other: Free Water Infusion

INTERVENTIONS:
Other: Enteral Dextrose Infusion — A standard solution of 50% Dextrose (0.85 kcal/mL) will be infused via enteral route at a rate of 10 mL per hour for a duration of 24 hours.
  Arms: Enteral Dextrose Infusion
Other: Free Water Infusion — An infusion of free water will be initiated via enteral route at a rate of 10 mL per hour for a duration of 24 hours.
  Arms: Placebo

SUMMARY:
This study is a prospective single-center randomized double-blinded placebo-controlled clinical trial testing the effects of early enteral dextrose as a therapeutic agent in critically ill patients with sepsis. Primary outcomes are differences in circulating plasma levels of the pro-inflammatory cytokine IL-6 to be tested 24 hours after the start of enteral infusion. Secondary outcomes include differences in circulating incretin hormone levels, differences in other pro-inflammatory cytokines including IL-1β and TNF-α, changes in intestinal microbial composition and function after intervention, glycemic control and variability as assessed by capillary blood glucose measurements and exogenous insulin dosing during the intervention period, and clinical outcomes including intensive care unit (ICU) and hospital stay and in-hospital mortality.

DETAILED DESCRIPTION:
The central objective of this research project is to determine how early caloric support impacts inflammatory and metabolic outcomes in the acute phase of sepsis. Preliminary data from our mouse models suggest that provision of dextrose via an intravenous route, even at low levels early in the course of sepsis, markedly impairs glucose tolerance and decreases insulin sensitivity and insulin secretion. In contrast, provision of low-level dextrose by the enteral route at identical levels during the early phase of sepsis is associated with decreased inflammation, increased secretion of beneficial intestine-derived incretin hormones, and significant improvements in glucose metabolism. The goals of this clinical study are to translate findings on the beneficial role of early enteral dextrose in a pilot interventional trial in critically-ill patients with sepsis. This clinical trial will provide further insight into the optimal timing and route of early caloric support in the care of septic patients-an area of clinical practice that will benefit from further studies in fundamental biology and clear guidelines for physicians.

ELIGIBILITY:
Inclusion Criteria:

1. New presentation of sepsis characterized by a confirmed or suspected infection, with an acute increase from baseline in a modified Sepsis-Related Organ Failure Assessment (SOFA) score of greater than or equal to 2 points. If baseline values are unknown, baseline SOFA score of 0 will be assumed.
2. Available enteral access defined by: (1) an existing nasogastric or orogastric tube, (2) plans to place a nasogastric or orogastric tube, or (3) an existing percutaneous endoscopic gastrostomy (PEG) tube.
3. Less than 48 hours since meeting criteria for sepsis.
4. Expected to stay at least 24 hours in the ICU.

Exclusion Criteria:

1. Pre-existing continuous enteral tube feed use prior to study entry.
2. Diabetic ketoacidosis or diabetic hyperosmolar hyperglycemic syndrome.
3. Previously enrolled in this study within the same hospital admission.
4. ICU physician request to exclude patient based on clinical assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Plasma IL-6 | 24 hours after start of infusion
  Pro-inflammatory cytokine

SECONDARY OUTCOMES:
Additional pro-inflammatory cytokines | 24 hours after start of infusion
  Circulating levels of other pro-inflammatory cytokines including IL-1 beta and TNF-alpha (each to be determined in pg/mL)
Incretin hormone levels | 24 hours after start of infusion
  Circulating levels of the intestine-derived hormones GIP and GLP-1 (each to be determined in pg/mL)
Microbiome composition | 24 hours after start of infusion
  Analysis of the composition and distribution of microorganisms of the gut and respiratory microbiome measured after intervention from tracheal aspirates and rectal swabs
Glycemic control | First 24 hours
  Capillary blood glucose measurements during infusion period
Mortality | 30 days
  In-hospital mortality at 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Faraaz A Shah, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shah FA, Kitsios GD, Yende S, Dunlap DG, Scholl D, Chuan B, Al-Yousif N, Zhang Y, Nouraie SM, Morris A, Huang DT, O'Donnell CP, McVerry BJ. A Pilot Double-Blind Placebo-Controlled Randomized Clinical Trial to Investigate the Effects of Early Enteral Nutrients in Sepsis. Crit Care Explor. 2021 Oct 8;3(10):e550. doi: 10.1097/CCE.0000000000000550. eCollection 2021 Oct. PMID 34651137
- [Derived] Shah FA, Mahmud H, Gallego-Martin T, Jurczak MJ, O'Donnell CP, McVerry BJ. Therapeutic Effects of Endogenous Incretin Hormones and Exogenous Incretin-Based Medications in Sepsis. J Clin Endocrinol Metab. 2019 Nov 1;104(11):5274-5284. doi: 10.1210/jc.2019-00296. PMID 31216011

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-24): https://cdn.clinicaltrials.gov/large-docs/87/NCT03454087/Prot_SAP_002.pdf